## UNIVERSIDAD NACIONAL AUTÓNOMA DE MÉXICO





## INFORMED CONSENT FORM

## Effect of dietary iodine supplementation on breast cancer proliferation

| Name of the patient |
|------------------------|
| Hospital |
| Responsible oncologist |

- I who subscribe, oncology patient, confirm that I have been invited to participate voluntarily in the clinical trial.
- I confirm that the medical staff or researcher has explained to me the characteristics of the trial, the iodine solution, its nature and the objectives of the study.
- I am aware that the protocol includes a group that will receive a solution without iodine (placebo), which will be the control group, and that I might belong to it.
- I am aware that 1% of people who take excess iodine can have side effects: stomach irritation, hives and / or acne.
- I am aware that I can leave the study freely after a simple notification and without detriment to my oncological treatment.
- I am aware that if iodine supplementation is beneficial, I can receive it for the first time (placebo group) or continue to receive it (iodine group) for free during my second period of chemotherapy.
- I confirm that I directly or through my legal representative have freely agreed to participate, signing this consent form along with two witnesses that I chose.
- I am aware that this document will be archived in the researchers' collection, where it will remain for at least 5 years after the end of the study.

| Signature of the patient/legal representative |
|-----------------------------------------------|
| Name and signature of witness 2 |

Instituto de Neurobiología, UNAM

Blvd. Juriquilla 3001

Juriquilla, Querétaro 76230